CLINICAL TRIAL: NCT06486740
Title: An Open-label Uncontrolled Single Centre Investigation for the Evaluation of the Safety and Performance Characteristics of the Dermal Filler, of Hyaluronic Acid 20 mg/ml, (M-AOX-2021) for Soft Tissue Augmentation Intended to be Used as a Temporary Dermal Filler for the Correction of Mild and Moderate Facial Wrinkles.
Brief Title: Evaluation of the Safety and Performance Characteristics of Mesofiller Aox for the Correction of Mild and Moderate Facial Wrinkles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mesoestetic Pharma Group S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-AOX-2021
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Skin Aging; Skin Wrinkling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesofiller aox (Experimental): The investigated product M-AOX-2021 was applied by intradermal or subcutaneous injection by the investigator during Session 1 for all subjects and Session 2 for the subjects, for whom a touch-up was considered beneficial. The both sessions was conducted within 14 days interval.
  Interventions: Device: mesofiller aox

INTERVENTIONS:
Device: mesofiller aox — The investigated product M-AOX-2021 was applied by intradermal or subcutaneous injection by the investigator during Session 1 for all subjects and Session 2 for the subjects, for whom a touch-up was considered beneficial. The both sessions was conducted within 14 days interval.

SUMMARY:
The investigation is a single centre, interventional, prospective, non-randomized, open-label, uncontrolled, single arm, un-blinded investigation for evaluation of safety and performance of the medical device M-AOX-2021 in the treatment of wrinkles and imperfections. The clinical investigation is interventional and prospective in agreement with the pre-market regulatory status of the product.

DETAILED DESCRIPTION:
The product M-AOX-2021 is a dermal filler manufactured by mesoestetic Pharma Group s.l.. It was intended to be used as a temporary dermal filler for dermatological treatment for aesthetic purposes. The product corrects wrinkles and imperfections of the lower two thirds of the face, while also providing hydration and an antioxidant action to the skin.

Мesofiller aox for facial area is a sterile, injectable, gel colourless, transparent, non-pyrogenic, reabsorbable medical device made out of cross-linked hyaluronic acid of non-animal origin, produced via bacterial fermentation.

This clinical investigation was conducted as an uncontrolled - no comparator medical device or other product was used. The safety and performance of the treatment was evaluated by comparison of the condition with the state of the treated area before initiation of the procedure, conducted by the trained Principal Investigator.

The investigated product M-AOX-2021 was applied by intradermal or subcutaneous injection by the investigator during Session 1 for all subjects and Session 2 for the subjects, for whom a touch-up was considered beneficial. The both sessions was conducted within 14 days interval.

The process of the evaluation during the medical examination was facilitated by photographic evidence taken before and after therapy at a predetermined time points for reference.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥20 and ≤70 years;
* Subjects presenting signs of skin depressions, scars or wrinkles in the lower two thirds of the face;
* Aesthetic scores of 2, 3 or 4 (mild, moderate or substantial loss of midface fullness, respectively) on each side of the face assessed at baseline by the investigator;
* Subject who is willing to abstain from any other facial aesthetic or cosmetic procedure or plastic surgery during the clinical investigation, including follow-up period;
* Subject who understands and is willing to comply with all investigation-related activities and who is available for the duration of their participation in the investigation, including follow-up;
* Absence of a history of significant hypersensitivity to food and drugs or known sensitivity to hyaluronic acid, lidocaine or other anesthetics or nerve-blocking agents;
* Arterial blood pressure (BP) (after 5 min. at rest in the supine position) in reference range - systolic 90 - 140 mmHg and diastolic 50 - 90 mmHg;
* Heart rate (HR) (after 5 min. at rest in the supine position) in reference range - over 50 beats/min and less than 100 beats/min;
* Axillar body temperature of up to 37°С;
* Clinical-laboratory examinations within the reference ranges or with no clinically significant abnormalities for CBC, ESR, PT/INR;
* Negative pregnancy test for the women with reproductive potential;
* Reliable and acceptable method of contraception for the women of child-bearing potential:

  * IUD, inserted at least 3 months prior to the investigation initiation;
  * Double barrier method (condom, spermicide-containing diaphragm) applied at least 14 days prior to the first investigated product application and throughout the course of the investigation;
  * Hormonal contraception with use initiation at least 3 months prior to the first investigated product application and throughout the course of the investigation;
  * Sexual abstinence for at least 14 days prior to enrollment into the investigation and throughout the course of the investigation;
  * Surgical sterilisation (bilateral ligation of the uterine tubes, hysterectomy, bilateral ovariectomy or vasectomy of the regular partner) with no less than a 6-month history;
  * Menopause with no less than a 2-year history prior to the investigation initiation.
* Signed written Informed Consent Form by the adult participant.

Exclusion Criteria:

* Subject with known severe or multiple allergies, including allergy or hypersensitivity to any of the DF components (HA, lidocaine, succinic acid, ascorbyl glucoside, idebenone) or other anesthetics or nerve-blocking agents,or significant allergy or hypersensitivity to food and drugs;
* History of any disease resulting in changes of facial contour or oedema of the face during the clinical investigation period;
* Ascertained tendency to develop hypertrophic or keloid scars or pigmentation disorders;
* History of connective tissues diseases;
* History of active autoimmune diseases or those under immunotherapy;
* History of or laboratory results suggesting coagulation disorder;
* Active skin disease or inflammation of or near the injection area that could interfere with the clinical investigation injections or assessments;
* Subject who suffers from another medical condition or who is receiving medication that in the Principal Investigator's judgment would prohibit inclusion in this investigation;
* Soft tissue augmentation with bovine collagen (in the previous 6 months), with porcine or human collagen (in the previous 12 months), or with hyaluronic acid or hydroxyapatite (in the previous 18 months);
* Subject with permanent implants in the neck or face within the previous 36 months;
* Any aesthetic treatment/procedure of the face in the previous 6 months that may interfere with the investigation's injections and/or investigation assessments, as judged by the investigator;
* Presence of any condition, which in the opinion of the investigator, makes the subject unable to complete the clinical investigation as per this CIP;
* Subject who is currently participating in another clinical investigation which may interfere with this clinical investigation results or who had participated in another clinical investigation within 30 days prior to enrollment in this investigation;
* Pregnancy, postpartum period (6 months), lactation or post-lactation period (6 months) or woman who plans pregnancy during the investigation follow-up period;
* Absence of a reliable and effective method of contraception for subject with childbearing potential;
* Known abuse of drugs, alcohol or other substances;
* Subject with limited mental and consistent comprehension abilities; incapacitated subjects; sportsmen and individuals on strenuous physical loading; prisoners;
* Refusal to sign the Informed Consent Form by the adult participant.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs, SAEs, ISRs, TEAEs | Two months after the first treatment (Session 3 (Day 60))

SECONDARY OUTCOMES:
Modified Fitzpatrick Wrinkle Scale (MFWS) - principal investigator evaluation. | Session 1 (Day 1), Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365).
  The absolute change in Modified Fitzpatrick Wrinkle Scale (MFWS) from baseline evaluated by the principal investigator based on the photographs of the treated area. MFWS is a wrinkle-scoring system for perioral and periorbital wrinkle severity, ranging from Class 1 Class 1 - mild to Class 3 - severe.
Modified Fitzpatrick Wrinkle Scale (MFWS) - patient evaluation. | Session 1 (Day 1), Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365).
  The absolute change in Modified Fitzpatrick Wrinkle Scale (MFWS) from baseline evaluated by the patient. MFWS is a wrinkle-scoring system for perioral and periorbital wrinkle severity, ranging from Class 1 Class 1 - mild to Class 3 - severe.
Global Aesthetic Improvement Scale (GAIS) - principal investigator evaluation. | Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365)
  Improvement in the Global Aesthetic Improvement Scale as evaluated by the principal investigator based on the photographs of the treated area. GAIS ranges from grade 1 to 5, where grade 1 shows exceptional improvement.
Global Aesthetic Improvement Scale (GAIS) - patient evaluation. | Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365)
  Improvement in the Global Aesthetic Improvement Scale as evaluated by the patient. GAIS ranges from grade 1 to 5, where grade 1 shows exceptional improvement.
Visual Analogous Scale (VAS) - principal investigator evaluation. | Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365)
  The absolute change in the Visual Analogous Scale from baseline judged by the principal investigator. VAS ranges from grade 0 to 10, where grade 10 is the best possible outcome.
Visual Analogous Scale (VAS) - patient evaluation | Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365)
  The absolute change in the Visual Analogous Scale from baseline judged by the patient. VAS ranges from grade 0 to 10, where grade 10 is the best possible outcome.
Subject satisfaction | Session 1 (Day 1), Session 2 (Day 14), Session 3 (Day 60), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365)
  The Patient's Questionnaire was utilised. The satisfaction survey grades range from 1 to 3, where grade 1 represents the highest satisfaction level.
Frequency and severity of AEs, SAEs, ISRs, TEAEs | Session 1 (Day 1), Session 2 (Day 14), Session 4 (Day 180), Session 5 (Day 270), and Session 6 (Day 365)

CONTACTS AND LOCATIONS:
Locations (1):
- "Medical Center Ramus" EOOD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No